CLINICAL TRIAL: NCT07078370
Title: Safety Study of Vascudyne's Small Diameter Acellular Tissue Engineered Vessel (ATEV) for Coronary Artery Bypass
Brief Title: Safety Study of Acellular Tissue Engineered Vessel for Coronary Artery Bypass
Acronym: VCAB-2
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Vascudyne, Inc. (Industry)
Collaborators: KCRI (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-004
Record Dates: First submitted 2025-06-29; First posted 2025-07-22 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease; Multi Vessel Coronary Artery Disease
Keywords: CABG; ATEV; Tissue Engineered Vessel; coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Patients will be implanted with a single Acellular Tissue Engineered Vessel with External Support Structure bypass (single proximal and distal anastomoses) to the second or third coronary artery bypass target
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- ATEV with ESS (Experimental): Surgical implant of Acellular Tissue Engineered Vessel with External Support Structure as Coronary Artery bypass
  Interventions: Device: ATEV with ESS

INTERVENTIONS:
Device: ATEV with ESS — Patients will be implanted with a single Acellular Tissue Engineered Vessel with External Support Structure bypass (single proximal and distal anastomoses) to the second or third coronary artery bypass target
  Other Names: CABG

SUMMARY:
To assess safety and feasibility of a coronary bypass created with Vascudyne Acellular Tissue Engineered Vessel (ATEV) with External Support Structure (ESS) in patients requiring multi vessel coronary artery bypass grafting (CABG).

DETAILED DESCRIPTION:
Prospective, non-randomized, evaluation clinical study to assess the feasibility of Acellular Tissue Engineered Vessel (ATEV) with External Support Structure (ESS) for secondary coronary targets in patients needing multiple coronary artery bypass.

Patients will be implanted with a single ATEV with ESS bypass (single proximal and distal anastomoses) to the second or third coronary arteries (CA) bypass target.

The primary target CA shall be bypassed using an arterial graft. The left anterior descending (LAD) CA bypass, if needed, shall be bypassed using the left internal mammary artery (LIMA). A native vessel shall be used for any additional targets as needed.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet ALL of the following inclusion criteria:

1. Patient with limited quantity of good quality saphenous vein graft (SVG) for planned operation per the surgeon discretion.
2. Bypass to at least three coronary arteries (CA); primary target shall be an Interior mesenteric artery (IMA) bypass to the Left anterior descending (LAD) artery, at least one SVG to a secondary CA target, and one Acellular Tissue Engineered Vessel (ATEV) to a secondary target CA that:

   * requires ≤ 15cm long conduit
   * has a diameter at least 1.5 mm at targeted landing site
   * has at least 70% stenosis proximal to the target bypass
   * has at least Thrombolysis in Myocardial Infarction (TIMI) flow grade II
3. Male or female patients between the ages of 45 and 75 years inclusive.
4. Elective patient, selected and accepted by the local Heart Team and confirmed by the Sponsor's Screening Committee for an on-pump full sternotomy coronary artery bypass grafting (CABG) surgery.
5. Concomitant life-threatening disease likely to limit life expectancy to less than 2 years.
6. Female subjects must be of non-childbearing potential, which is defined as post-menopausal (at least 1 year without menses prior to Screening) or documented surgically sterile or post hysterectomy (at least 1 month prior to Screening).
7. Patient has been informed of the nature of the study, agrees to its provisions, and has provided written informed consent.
8. Patient has been informed and agrees to pre- and post-procedure follow-up, including follow-up cardiac ultrasound and coronary angiogram or computed tomography (CT).
9. Patient is willing to be compliant with prescribed anticoagulant therapy (critical to preventing thrombus in the ATEV).

Exclusion Criteria:

1. Patients with left ventricular ejection fraction < 35%.
2. Patients with diffusely diseased coronary arteries suggestive of either poor target quality, or poor vessel runoff.
3. Patients requiring emergency surgery.
4. Patients with cardiogenic shock.
5. Patients with any prior open cardiac surgery such as CABG.
6. Any planned concomitant cardiac surgery, including but not limited to: valve surgery, repair of intracardiac shunt, surgical arrhythmia ablation.
7. History of cardiac resynchronization therapy (CRT) or implantable cardioverter defibrillator (ICD) implantation.
8. Myocardial infarction (MI) within 21 days or cerebral vascular accident (CVA) within 90 days of the CABG procedure.
9. Patient with uncontrolled diabetes (glycated hemoglobin > 8%).
10. Chronic Kidney Disease (CKD) with Glomerular Filtration Rate (GFR) <45 mL/min/1.73m2 (Category: G3b-G5 according to Kidney Disease: Improving Global Outcomes (KDIGO)).
11. Moderate to severe chronic obstructive pulmonary disease (COPD) with a forced expiratory volume (FEV) <1.5 L/sec or 45% predicted FEV1.
12. Patient with known interstitial lung disease, diagnosed by imaging or pulmonary function tests, including Diffusing Capacity of the Lungs for Carbon Monoxide (DLCO).
13. Endocarditis, pericarditis, or any other active systemic infection that would interfere with patient safety.
14. Patient on preoperative anticoagulant, or pre existing indication for anticoagulation (e.g. atrial fibrillation, history of thromboembolism), or with known coagulation disorder.
15. Abnormal blood values (e.g. leukopenia, anemia, thrombocytopenia, or thrombocytosis with Platelet Count >400,000 per mL that could influence graft hemostasis or patient recovery
16. Known allergies to study device components: Nitinol, Nickel, Titanium, or agents/medication such as contrast agents, antiplatelet therapy, beta-blocker, or statins required for study assessment or optimal post-CABG medical treatment (hospital standard of care).
17. Contraindication to or known serious allergy to anticoagulant, aspirin, or planned antiplatelet (clopidogrel, ticagrelor, prasugrel) and factor Xa inhibitor therapy.
18. Any planned medical intervention or condition within the 12 months following ATEV implantation that requires temporary or permanent discontinuation of antiplatelet or anticoagulant therapy.
19. History of heparin-induced thrombocytopenia.
20. Documented or suspected untreated diffuse peripheral vascular disease such as: carotid stenosis or claudication of the extremities.
21. Immunodeficiency including Human Immunodeficiency Virus (HIV), active autoimmune disease, or on immunosuppressant therapy.
22. Treatment with any investigational drug or device within 60 days prior to study entry or ongoing participation in another clinical study of an investigational product.
23. Subject has medical, social, or psychosocial factors that, in the opinion of the investigator, could impact safety or compliance.
24. Has any other condition, in the opinion of the principal investigator, which would put the patient at increased risk from participating in the study or otherwise prevent participation.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Successful implantation | 30 days.
  Successful implantation as defined by meeting each of the following points:
  1. Completion of both a proximal and distal anastomosis,
  2. Placement of ESS,
  3. No evidence of ATEV twist or kink on direct visual inspection.
Freedom from Major Adverse Cardiac and Cerebrovascular events (MACCE) at 30 days. | 30 days.
  Freedom from Major Adverse Cardiac and Cerebrovascular events (MACCE) at 30 days. MACCE is defined as combination of:
  1. death,
  2. non-fatal stroke,
  3. non-fatal myocardial infarction,
  4. unplanned revascularization
  5. hospitalization due to heart failure

SECONDARY OUTCOMES:
Patency at 1 and 6 months | 1 month and 6 months.
  Patency of conduit assessed by Coronary Computed Tomography Angiography (CCTA) results at 1 and 6 months post-implantation.
Patency at 12 months | 12 months.
  Patency of conduit assessed by angiography results at 12 months, defined according to Fitzgibbon classification.
Lumen Diameter Uniformity | 12 months.
  Lumen Diameter Uniformity of all bypasses assessed by angiography results at 12 months.
Immune Response | 12 months.
  Panel Reactive Antibody assessment via serum assay at baseline, 1, 6, and 12 months.
Device Serious Adverse Event (SAE) | 6 months, 12 months, 24 months, 48 months, and 60 months.
  Device Related Serious Adverse Events identified at 6, 12, 24, 48 and 60 months follow-ups.
Freedom from (major adverse cardiac and cerebrovascular events) MACCE | 6 months, 12 months, 24 months, 48 months, and 60 months.
  Freedom from (major adverse cardiac and cerebrovascular events) MACCE at 6, 12, 24, 48 and 60 months follow-ups.

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof Wrobel, MD PhD, Principal Investigator — MEDICOVER SP Z O.O.
Locations (2):
- Poland (2):
  - University Clinical Hospital No. 2 PUM in Szczecin, Szczecin
  - Medicover, Warsaw

IPD SHARING:
Plan to Share IPD: No